CLINICAL TRIAL: NCT05114343
Title: Effectiveness and Feasibility of a Technology-supported Home-based Exercise Program for Adolescents With Juvenile Idiopathic Arthritis (THE_JIA Study): a Randomized Controlled Trial.
Brief Title: Effectiveness and Feasibility of a Home-based Exercise Program for Adolescents With Juvenile Idiopathic Arthritis
Acronym: THE_JIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: THE_JIA study
Record Dates: First submitted 2021-10-07; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-08

CONDITIONS: Juvenile Idiopathic Arthritis; Juvenile Arthritis; Juvenile Rheumatoid Arthritis
Keywords: physical activity; exercise; vascular function; endothelial function; feasibility; home-based exercise
MeSH Terms: conditions — Arthritis, Juvenile; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Primary outcome (i.e., endothelial function) will be assessed by a blinded investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Participants will be instructed to perform 3 sessions of weight-bearing exercise per week, for 12 weeks. Exercise intensity and duration will be low-to-moderate in the first 4 weeks, and will progressively increase during the program. Participants will be supported by educational materials, a heart rate monitor, and by means of periodic contact with an exercise specialist via video and phone calls, and text messages.
  Interventions: Behavioral: Exercise
- Usual care (control group) (No Intervention): Participants in the control group will receive usual care and general instructions about physical activity.

INTERVENTIONS:
Behavioral: Exercise — Participants will perform weight-bearing exercises for 12 weeks. The intervention will be delivered remotely through video calling with an exercise specialist.
  Other Names: physical activity
  Arms: Exercise group

SUMMARY:
This study will aim to test the effectiveness and feasibility of a technology-supported home-based exercise program in adolescents with JIA. For this, adolescents (< 18 years) with JIA will be randomized to a 12-weeks home-based exercise program or usual care (i.e., no exercise control intervention). The home-based exercise intervention will be delivered remotely using a video calling app, and participants will be instructed to perform 3 sessions of weight-bearing exercise per week. Participants will be supported by educational materials, a heart rate monitor, and through periodic contact with an exercise specialist via video and phone calls, and text messages. The study's primary outcomes will be: cardiac and vascular function and structure using ultrasound imaging, body composition (DXA), aerobic capacity, muscle strength and functional capacity. In addition to that, the feasibility, safety, acceptability, and barriers and facilitators to the intervention will also be assessed.

DETAILED DESCRIPTION:
Juvenile idiopathic arthritis (JIA) is the most common type of arthritis in children and adolescents under the age of 16. In addition to the articular features of the disease, JIA is also characterized by multiple comorbidities, including cardiovascular manifestations. Part of the health conditions observed in adolescents with JIA may be caused by a reduced practice of physical activity. Lack of physical activity in this disease has been attributed to generic and specific barriers, such as time constraints, low motivation, limited access to specialized exercise centers, lack of specific programs for JIA patients, among others. More recently, the COVID-19 pandemic has imposed additional challenges for the engagement in physical activity in populations with chronic disease, including patients with JIA. In this scenario, home-based exercise programs supported by technology have arisen as potentially effective alternatives to upregulate physical activity levels in adolescents with JIA, which needs to be further explored. Therefore, the aim of this study will be to test the effectiveness and feasibility of a technology-supported home-based exercise program in adolescents with JIA. For this, adolescent (< 18 years) patients with JIA will be randomized to a 12-weeks home-based exercise program or usual care (i.e., no exercise control intervention). The home-based exercise intervention will be delivered remotely using a video calling app, and participants will be instructed to perform 3 sessions of weight-bearing exercise per week. Exercise intensity and duration will be low-to-moderate in the first 4 weeks, and will progressively increase during the program. Participants will be supported by educational materials, a heart rate monitor, and by means of periodic contact with an exercise specialist via video and phone calls, and text messages. Participants in the control group will receive usual care and general instructions about physical activity. The study's primary outcome will be the cardiac and vascular structure and function assessed by vascular ultrasound imaging, body composition (DXA), aerobic capacity, muscle strength and functional capacity. Secondary outcomes will include clinical aspects of the disease, blood parameters, physical activity and sedentary behavior, food consumption, health-related quality of life, blood pressure, and cardiac autonomic function. Feasibility, safety, acceptability, and barriers and facilitators to the intervention will also be evaluated. The effects of the intervention on study outcomes will be assessed by a mixed model analysis (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Patients with polyarticular or oligoarticular subtypes of juvenile idiopathic arthritis.

Exclusion Criteria:

* Cardiovascular, metabolic, pulmonary or renal diseases
* Untreat thyroid disease
* Blood pressure > 140/80 mmHg
* Use of statin
* Use of tobacco
* Any other disease or condition that may prevent the practice of physical activity

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Endothelial function | Change from baseline to 12 weeks
  Endothelial function will be assessed through the evaluation of brachial flow-mediated dilation using a vascular ultrasound.
Cardiac chamber dimensions (left ventricle diastolic and systolic diameters, interventricular septum, left ventricular posterior wall) | Change from baseline to 12 weeks
  Left ventricle diastolic and systolic diameters, interventricular septum, and left ventricular posterior wall in millimeters per meter squared will be assessed using standard echocardiography.
Left ventricular ejection fraction (LVEF) | Change from baseline to 12 weeks
  Left ventricular ejection fraction (LVEF) in percentage will be assessed using standard echocardiography.
Left ventricular mass index | Change from baseline to 12 weeks
  The left ventricular mass index in grams per body surface area will be assessed using standard echocardiography.
Left ventricular diastolic function | Change from baseline to 12 weeks
  Left ventricular diastolic function will be assessed using tissue Doppler-based measurements of transmitral E and A velocities in metre per second.
Myocardial deformation | Change from baseline to 12 weeks
  Myocardial deformation in longitudinal, radial, and circumferential directions will be assessed using two-dimensional speckle-tracking (2DST) echocardiography and expressed as a percentage.
Body fat | Change from baseline to 12 weeks
  Body fat in % will be assessed using dual-energy X-ray absorptiometry.
Lean mass | Change from baseline to 12 weeks
  Lean mass in kilograms will be assessed using dual-energy X-ray absorptiometry.
Bone mineral content | Change from baseline to 12 weeks
  Bone mineral content in grams will be assessed using dual-energy X-ray absorptiometry.
Aerobic fitness | Change from baseline to 12 weeks
  Aerobic fitness will be assessed through a graded treadmill exercise test. VO2max will be assessed using a metabolic cart and expressed in millilitres per kilograms of body weight.
Vascular structure | Change from baseline to 12 weeks
  Vascular structure will be assessed through the analysis of common carotid intima-media thickness using a vascular ultrasound.
Feasibility of the intervention | Change from baseline to 12 weeks
  Feasibility of the intervention will be assessed through interviews investigating the experiences of the participants during the intervention.
Adherence to the intervention | Change from baseline to 12 weeks
  The adherence to the intervention will be assessed using the data from the physical activity diaries and heart rate monitor and will be expressed as percentage of complete sessions.

SECONDARY OUTCOMES:
Disease activity | Change from baseline to 12 weeks
  Participants' disease activity will be calculated using the Juvenile Arthritis Disease Activity Score.
Disease activity | Change from baseline to 24 weeks
  Participants' disease activity will be calculated using the Juvenile Arthritis Disease Activity Score.
Functional ability | Change from baseline to 12 weeks
  The functional ability of the participants with JIA will be assessed through the Brazilian-Portuguese version of the Childhood Health Assessment Questionnaire (CHAQ).
Functional ability | Change from baseline to 24 weeks
  The functional ability of the participants with JIA will be assessed through the Brazilian-Portuguese version of the Childhood Health Assessment Questionnaire (CHAQ).
Health-related quality of life | Change from baseline to 12 weeks
  Health-related quality of life will be assessed through the Pediatric Quality of Life Inventory (PedsQL).
Health-related quality of life | Change from baseline to 24 weeks
  Health-related quality of life will be assessed through the Pediatric Quality of Life Inventory (PedsQL).
Cardiometabolic blood markers | Change from baseline to 12 weeks
  The following cardiometabolic markers from blood will be assessed after 12-h fasting: blood glucose and insulin, total cholesterol, HDL cholesterol, LDL cholesterol, VLDL cholesterol, and triglycerides. This data will be expressed in milligrams per deciliter.
C-reactive protein | Change from baseline to 12 weeks
  C-reactive protein levels in the blood will be assessed after 12-h fasting and expressed as milligrams per litre.
Physical activity and sedentary behavior | Change from baseline to 12 weeks
  Physical activity and sedentary behavior will be assessed using a thigh-worn accelerometer (activPAL).
Physical activity and sedentary behavior | Change from baseline to 24 weeks
  Physical activity and sedentary behavior will be assessed using a thigh-worn accelerometer (activPAL).
Motivation to physical activity | Change from baseline to 12 weeks
  Motivation to physical activity will be assessed using the Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2).
Physical activity-related behavior | Change from baseline to 12 weeks
  Physical activity-related behavior will be asseessed using the Stages of Change model.
Food consumption | Change from baseline to 12 weeks
  Food consumption will be assessed through 24-hour food recalls, collected on three non-consecutive days (one weekend day).
Blood pressure | Change from baseline to 12 weeks
  Blood pressure (arterial pressure) will be assessed non-invasively using a multi-parameter monitor.
Cardiac autonomic function | Change from baseline to 12 weeks
  Cardiac autonomic function will be assessed through the analysis of heart rate variability, which will be recorded using a heart rate monitor.
Muscle strength | Change from baseline to 12 weeks
  Muscle strength will be assessed by the one-repetition maximum test on the bench press and knee extension machines and will be expressed as kilograms.
Muscle strength | Change from baseline to 24 weeks
  Muscle strength will be assessed by the one-repetition maximum test on the bench press and knee extension machines and will be expressed as kilograms.
Handgrip strength | Change from baseline to 12 weeks
  Handgrip strength will be assessed using handgrip dynamometry and expressed as kilograms.
Handgrip strength | Change from baseline to 24 weeks
  Handgrip strength will be assessed using handgrip dynamometry and expressed as kilograms.
Functional capacity - Timed-Stands | Change from baseline to 12 weeks
  Functional capacity will be assessed using the "Timed-Stands" test and expressed by the number of sit-to-stand repetitions.
Functional capacity - Timed-Stands | Change from baseline to 24 weeks
  Functional capacity will be assessed using the "Timed-Stands" test and expressed by the number of sit-to-stand repetitions.
Functional capacity - Timed Up-And-Go | Change from baseline to 12 weeks
  Functional capacity will be assessed busing the "Timed Up-And-Go" test and expressed in seconds.
Functional capacity - Timed Up-And-Go | Change from baseline to 24 weeks
  Functional capacity will be assessed busing the "Timed Up-And-Go" test and expressed in seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da USP - HCFMUSP, São Paulo, Brazil